CLINICAL TRIAL: NCT04565821
Title: Feasibility Study to Assess a Trans-nasal Intestinal Potential Difference Probe
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator - MD, PhD, FACC, FCAP, FNAI, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2020P000158
Record Dates: First submitted 2020-08-11; First posted 2020-09-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Disease; Permeability; Increased; Crohn Disease; Inflammatory Bowel Diseases; Environmental Enteropathy
Keywords: OCT; Optical Coherence Tomography; TNIT; Trans Nasal Introduction Tube; IPD; Intestinal Potential Difference; Leaky Gut; Gastrointestinal Permeability; GI Permeability
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Feasibility of trans-nasal IPD probe (Experimental): The purpose of this study is to examine the feasibility of using a trans-nasal IPD probe as a measurement tool for gut permeability
  Interventions: Device: IPD Probe via TNIT

INTERVENTIONS:
Device: IPD Probe via TNIT — A total of 10 healthy adult volunteers will be enrolled in this study. All consented participants will be receive the same intervention. A Nasal tube will be inserted through nares until reaching the small intestine. This will be confirmed by m-mode OCT. Once secured, we will start infusing Ionic solution into the intestine so that IPD Probe can measure the potential difference between this and the control reading. The control reading is measured by infusing the same ionic solution subcutaneously on large muscle groups.

SUMMARY:
The purpose of this study is to examine the feasibility of using a trans-nasal IPD probe as a measurement tool for gut permeability

DETAILED DESCRIPTION:
Increased gastrointestinal (GI) permeability is associated to several GI conditions that affect millions of people worldwide. Healthy intestinal walls limit only specific molecules to cross into the body. "Leaky gut" is a condition of unregulated and increased gut permeability that allows unwanted antigens, pathogens and microbial toxins into the bloodstream(1). This in turn leads to a subsequent immune response that includes the production of inflammatory mediators. Leaky gut is a key feature in celiac disease, Crohn's disease, inflammatory bowel disease (IBD), and environmental enteropathy and have been associated with systemic diseases including type 1 diabetes, autoimmune hepatitis, and systemic lupus erythematosus (SLE).

The current gold standard for measuring intestinal permeability is the sugar ratio test. Non-metabolized sugars of different molecular sizes are orally administered and the amount of sugar molecules absorbable across the gut lining is then quantified by measuring their relative concentrations in urine. In healthy subjects, low to none of the large-molecule disaccharides can be taken into the circulatory system, while the small-molecule monosaccharides can readily diffuse into the bloodstream. This results in low disaccharide/monosaccharide (DM) ratios for healthy subjects. Subjects with the leaky gut conditions exhibit high DM ratios in their urine. However, the sugar ratio test has low specificity, does not provide specific information on etiology, is challenging to implement when pristine urine samples cannot be collected (e.g. infants), and does not account for spatially heterogeneous disease.

An alternative approach for measuring mucosal permeability is through measuring the voltage across the intestinal wall (Intestinal potential difference; IPD) that changes with intestinal permeability. The Tearney lab has developed an IPD measuring device (IPD probe) that can be deployed trans-nasally and can measure the intestinal potential difference in real time at selected locations of the gut. The probe contains a central channel that allows us to infuse specific ionic solutions into the gut. The IPD probe also has an optical fiber inside the channel that enables the acquisition of M-mode OCT images. The M-mode OCT images make it possible to determine when the IPD probe is in contact with the tissue.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Participant must be 18 to 60 years of age
* Participant must be able to consent to the procedure
* Participant must fast (no solid food) for at least 8 hours prior to the procedure

Exclusion Criteria:

* Participants with a history of upper respiratory disease or surgery
* Participants with a history of upper gastrointestinal surgery
* Partcipants with upper respiratory infection at least 7 days prior to the procedure
* Participants with any contraindications to the placement of the NJ tube including deviated septum or any other anatomical abnormalities of the nasopharynx or upper gastrointestinal region, history of trans-sphenoidal surgery, facial or cranial trauma and fractures, chronic sinusitis, esophageal strictures, varices etc.
* Participants with a history of or being on medications that delay gastric emptying.
* Participants on drugs which impair clotting like anticoagulants and antiplatelet drugs, NSAIDS, history of bleeding disorders.
* Participants using nasal steroids or any steroids for environmental allergies
* Participants with suspected or diagnosed HIV
* Participants with a recent use of Antibiotics within the past 4 weeks
* Participants with a current or history of Alcoholism
* Participants with suspected or diagnosed Hep B or Hep C
* Participants enrolled in clinical trials involving interventions that affect Intestinal Permeability
* Participants with uncontrolled Diabetes Mellitus 1 & Diabetes Mellitus 2
* Participants currently taking H2 Histamine Antagonists (such as Pepcid, Axid, Tagamet, Zantac, etc)
* Participants currently taking Mast Cell stabilizers
* Participants currently pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Baseline IPD readings | The outcome measure is actively recorded in real-time during the procedure, an average of 3 hours.
  Feasibility will be measured by the IPD probes ability to, accurately and in real-time, measure voltages that are consistent with literature for the tissue we are testing
IPD readings after Glucose/Galactose infusion | The outcome measure is actively recorded in real-time during the procedure, an average of 3 hours.
  the IPD probe's ability to measure a more positive reading when Glucose or Galactose have been perfused.
Image Quality | Imaging data is collected during the procedure, and analyzed within 1 year of collection.
  Image quality will be determined by our study staff's ability to discern the various tissues' architecture and morphology and the resolution of the images recorded. This is a qualitative measurement to determine feasibility of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D, PhD., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No